CLINICAL TRIAL: NCT04509869
Title: Outcome of Subinguinal Varicocelectomy on Normal Semen in Patients Complaining of Orchialgia
Brief Title: "Outcome of Varicocelectomy on Normal Semen in Patients Complaining of Orchialgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Mohamed Abdelkader, chief resident of urology, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: orchialgia treatment
Record Dates: First submitted 2020-08-07; First posted 2020-08-12 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Varicocele; Pain; Fertility Issues
MeSH Terms: conditions — Varicocele; Pain; Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pre-operative and postoperative (Experimental): the patients who will undergo the operation to treat the pain
  Interventions: Procedure: varicocelectomy

INTERVENTIONS:
Procedure: varicocelectomy — operation for varix ligation

SUMMARY:
varicoclelectomy is done for subfertiltiy and varicocele induced orchialgia. The effect of varicocelectomy on semen analysis is controversial. Many articles report favorable outcomes and others do not.

Most study don't focus on varicocelectomy done for varicocele induced orchialgia,and those studies dont report on postoperative semen.

This study will focus on the effect of operation on the semen postoperatively .

ELIGIBILITY:
Inclusion Criteria:

1. Primary varicocele
2. Patient's age more than 19 years
3. Normal semen analysis (according to the WHO 5th guide to semen parameters where sperm concentration equal 15 million per ml , total sperm number 40 million per ejaculate ,normal morphology 4 % and motility A =25% or a+b = 32% is considered normal.
4. Scrotal pain after exclusion of other causes.

Exclusion Criteria:

* 1- Recurrent varicocele

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2017-08-12 (Actual); Primary Completion 2020-08-12 (Actual); Study Completion 2020-08-12 (Actual)

PRIMARY OUTCOMES:
sperm motility | 3 months postoperative is our aim
  semen analysis will be done preoperative and post-operative
sperm morphology | 3 months postoperative is our aim
  semen analysis will be done preoperative and postoperative
sperm number | 3 months postoperative is our aim
  semen analysis will be done preoperative and postoperative
pain of scrotum | 3 months postoperative is our aim
  subjective sensation measured by visual analogue score preoperative and postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Assuit Medical School, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chen SS. Factors predicting symptomatic relief by varicocelectomy in patients with normospermia and painful varicocele nonresponsive to conservative treatment. Urology. 2012 Sep;80(3):585-9. doi: 10.1016/j.urology.2012.05.014. Epub 2012 Jul 10. PMID 22784493
- [Background] Abd Ellatif ME, Asker W, Abbas A, Negm A, Al-Katary M, El-Kaffas H, Moatamed A. Varicocelectomy to treat pain, and predictors of success: a prospective study. Curr Urol. 2012 May;6(1):33-6. doi: 10.1159/000338867. Epub 2012 Mar 18. PMID 24917707
- [Background] Cho CL, Esteves SC, Agarwal A. Indications and outcomes of varicocele repair. Panminerva Med. 2019 Jun;61(2):152-163. doi: 10.23736/S0031-0808.18.03528-0. PMID 30990285
- [Background] Maghraby HA. Laparoscopic varicocelectomy for painful varicoceles: merits and outcomes. J Endourol. 2002 Mar;16(2):107-10. doi: 10.1089/089277902753619627. PMID 11962551
- [Background] Peterson AC, Lance RS, Ruiz HE. Outcomes of varicocele ligation done for pain. J Urol. 1998 May;159(5):1565-7. doi: 10.1097/00005392-199805000-00043. PMID 9554356
- [Background] Yaman O, Ozdiler E, Anafarta K, Gogus O. Effect of microsurgical subinguinal varicocele ligation to treat pain. Urology. 2000 Jan;55(1):107-8. doi: 10.1016/s0090-4295(99)00374-x. PMID 10654904